CLINICAL TRIAL: NCT02316353
Title: An Open-label, Randomized Study to Evaluate the Long-term Clinical Safety and Efficacy of Subcutaneous Administration of Human Plasma-derived C1-esterase Inhibitor in the Prophylactic Treatment of Hereditary Angioedema
Brief Title: A Study to Evaluate the Long-term Clinical Safety and Efficacy of Subcutaneously Administered C1-esterase Inhibitor in the Prevention of Hereditary Angioedema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSL830_3002; 2014-001054-42 (EudraCT Number)
Record Dates: First submitted 2014-12-10; First posted 2014-12-12 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2017-10

CONDITIONS: Hereditary Angioedema Types I and II
MeSH Terms: conditions — Hereditary Angioedema Types I and II | interventions — Complement C1 Inhibitor Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- C1-INH - low-volume dose (Experimental): A low-volume dose of C1-INH will be administered subcutaneously twice a week for up to 52 weeks (up to 146 weeks extension period).
  Interventions: Biological: C1-esterase inhibitor
- C1-INH - medium-volume dose (Experimental): A medium-volume dose of C1-INH will be administered subcutaneously twice a week for up to 52 weeks (up to 146 weeks extension period).
  Interventions: Biological: C1-esterase inhibitor

INTERVENTIONS:
Biological: C1-esterase inhibitor

SUMMARY:
The aim of this study is to assess the long-term safety of C1-esterase inhibitor (C1-INH) in preventing hereditary angioedema (HAE) attacks when it is administered under the skin of subjects with HAE. The safety of participating subjects will be assessed for up to 54 weeks. The long-term efficacy of C1-INH will also be assessed. Each eligible subject will enter the treatment phase, wherein subjects will be randomized to treatment with either low- or medium-volume C1-INH. Subjects who have an insufficient treatment response during the study will be given an opportunity to undergo a dose increase. The study aims to enroll eligible subjects who completed study CSL830_3001 (NCT01912456). Subjects who did not participate in study CSL830_3001 may also participate, if eligible and if space permits. Subjects from the United States (US) who complete Treatment Period 2 will be allowed to participate in an Extension Period. During the Extension Period participating US subjects will continue to receive treatment with open-label CSL830 for up to an additional 88 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 6 years or older.
* A confirmed diagnosis of HAE type I or II.
* HAE attacks over a consecutive 2-month period that required acute treatment, medical attention, or caused significant functional impairment.
* For subjects who have used oral therapy for prophylaxis against HAE attacks within 3 months of first study visit: use of a stable regimen within 3 months of the first study visit.

Exclusion Criteria:

* Incurable malignancies.
* Any clinical condition that will interfere with the evaluation of C1-INH therapy.
* Clinically significant history of poor response to C1-esterase therapy for the management of HAE.
* Suspected or confirmed diagnosis of acquired HAE or HAE with normal C1-INH.
* Inability to have HAE managed pharmacologically with on-demand treatment.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2014-12-31 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2017-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Program Director, Study Director — CSL Behring
Locations (31):
- United States (12):
  - Study Site, Birmingham, Alabama
  - Study Site, Scottsdale, Arizona
  - Study Site, La Jolla, California
  - Study Site, Orange, California
  - Study Site, Walnut Creek, California
  - Study Site, Chevy Chase, Maryland
  - Study Site, Cincinnati, Ohio
  - Study Site, Tulsa, Oklahoma
  - Study Site, Portland, Oregon
  - Study Site, Hershey, Pennsylvania
  - Study Site, Dallas, Texas
  - Study Site, Richmond, Virginia
- Study Site, Campbelltown, New South Wales, Australia
- Canada (4):
  - Study Site, Hamilton, Ontario
  - Study Site, Ottawa, Ontario
  - Study Site, Toronto, Ontario
  - Study Site, Québec
- Study Site, Pilsen, Czechia
- Germany (4):
  - Study Site, Mörfelden-Walldorf, Hesse
  - Study Site, Berlin
  - Study Site, Frankfurt
  - Study Site, Mainz
- Study Site, Budapest, Hungary
- Israel (2):
  - Study Site, Tel Aviv
  - Study Site, Tel Litwinsky
- Italy (2):
  - Study Site, Catania
  - Study Site, Milan
- Study Site, Cluj-Napoca, Romania
- Spain (2):
  - Study Site, Madrid
  - Study Site, Valencia
- Study Site, London, United Kingdom

REFERENCES:
- [Derived] Beard N, Frese M, Smertina E, Mere P, Katelaris C, Mills K. Interventions for the long-term prevention of hereditary angioedema attacks. Cochrane Database Syst Rev. 2022 Nov 3;11(11):CD013403. doi: 10.1002/14651858.CD013403.pub2. PMID 36326435
- [Derived] Lumry WR, Zuraw B, Cicardi M, Craig T, Anderson J, Banerji A, Bernstein JA, Caballero T, Farkas H, Gower RG, Keith PK, Levy DS, Li HH, Magerl M, Manning M, Riedl MA, Lawo JP, Prusty S, Machnig T, Longhurst H; on behalf of the COMPACT Investigators. Long-term health-related quality of life in patients treated with subcutaneous C1-inhibitor replacement therapy for the prevention of hereditary angioedema attacks: findings from the COMPACT open-label extension study. Orphanet J Rare Dis. 2021 Feb 15;16(1):86. doi: 10.1186/s13023-020-01658-4. PMID 33588897
- [Derived] Levy DS, Farkas H, Riedl MA, Hsu FI, Brooks JP, Cicardi M, Feuersenger H, Pragst I, Reshef A. Long-term efficacy and safety of subcutaneous C1-inhibitor in women with hereditary angioedema: subgroup analysis from an open-label extension of a phase 3 trial. Allergy Asthma Clin Immunol. 2020 Feb 4;16:8. doi: 10.1186/s13223-020-0409-3. eCollection 2020. PMID 32042283
- [Derived] Craig T, Zuraw B, Longhurst H, Cicardi M, Bork K, Grattan C, Katelaris C, Sussman G, Keith PK, Yang W, Hebert J, Hanzlikova J, Staubach-Renz P, Martinez-Saguer I, Magerl M, Aygoren-Pursun E, Farkas H, Reshef A, Kivity S, Neri S, Crisan I, Caballero T, Baeza ML, Hernandez MD, Li H, Lumry W, Bernstein JA, Hussain I, Anderson J, Schwartz LB, Jacobs J, Manning M, Levy D, Riedl M, Christiansen S, Feuersenger H, Pragst I, Mycroft S, Pawaskar D, Jacobs I; COMPACT Investigators. Long-Term Outcomes with Subcutaneous C1-Inhibitor Replacement Therapy for Prevention of Hereditary Angioedema Attacks. J Allergy Clin Immunol Pract. 2019 Jul-Aug;7(6):1793-1802.e2. doi: 10.1016/j.jaip.2019.01.054. Epub 2019 Feb 15. PMID 30772477

RESULTS

PARTICIPANT FLOW:
Groups:
- CSL830 (40): A low-volume dose of C1-INH (40 IU/kg) administered subcutaneously twice a week
- CSL830 (60): A high-volume dose of C1-INH (60 IU/kg) administered subcutaneously twice a week
Period: Overall Study
Arm/Group | CSL830 (40) | CSL830 (60)
Started | 63 (7 subjects assigned to the CSL830 (40) Arm, were titrated up to the 60 IU/kg arm during the study) | 63
Completed | 55 | 55
Not Completed | 8 | 8
Not completed — Pregnancy | 1 | 3
Not completed — Adverse Event | 1 | 3
Not completed — Withdrawal by Subject | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CSL830 (40) | CSL830 (60) | Total
Number analyzed (Participants) | 63 | 63 | 126
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 5 | 11
  Between 18 and 65 years | 55 | 50 | 105
  >=65 years | 2 | 8 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (14.96) | 40.3 (16.26) | 40.5 (15.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 36 | 76
  Male | 23 | 27 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 59 | 59 | 118
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 4 | 12
  Romania | 1 | 0 | 1
  Hungary | 1 | 5 | 6
  United States | 25 | 29 | 54
  Czechia | 2 | 2 | 4
  Italy | 3 | 1 | 4
  United Kingdom | 1 | 1 | 2
  Israel | 6 | 8 | 14
  Australia | 1 | 2 | 3
  Germany | 13 | 9 | 22
  Spain | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Person-time Incidence Rates (Subject Based)
Description: Subject-based Analysis for Person-Time Incidence Rate = (the total number of subjects who experienced the event during the respective treatment) / (the sum of the date each subject experienced the event - the subject's start date + 1 day) / (365.25 days). The analysis population for this endpoint was the Safety Population: the Safety Population comprised all subjects who provided informed consent / assent, who were randomized, and who received at least 1 dose or a partial dose of CSL830.
Time Frame: Up to 146 weeks.
Population: Safety population: The Safety Population comprised all subjects who provided informed consent / assent, who were randomized, and who received at least 1 dose or a partial dose of CSL830.
Measure: Number; unit: participants with events/year
Arm/Group | CSL830 (40) | CSL830 (60)
Number analyzed (Participants) | 63 | 70
participants with events/year
  AEs Leading to Premature Study Discontinuation | 0.01 | 0.03
  Thromboembolic Events | 0.00 | 0.01
  Anaphylaxis | 0.00 | 0.00
  HAE Attacks Resulting in In-Patient Hospitalizatio | 0.00 | 0.00
  Solicited AEs Graded as Severe | 0.00 | 0.00
  Related SAEs Other Than Specified Above | 0.00 | 0.00
  Antibodies to C1-INH (Inhibitory + Non-inhibitory) | 0.06 | 0.06

2. Primary Outcome: The Person-time Incidence Rates (Event Based)
Description: Event-based Analysis for Person-Time Incidence Rate = (the total number of events documented during the respective treatment) / (the sum of each subject's end date - the subject's start date + 1 day) / (365.25 days). The analysis population for this endpoint was the Safety Population: The Safety Population comprised all subjects who provided informed consent / assent, who were randomized, and who received at least 1 dose or a partial dose of CSL830.
Time Frame: Up to 146 weeks.
Population: as for outcome 1
Measure: Number; unit: events/year
Groups:
- CSL830 (60): A high-volume dose of C1-INH (60 IU/kg) administered subcutaneously twice a week. Actual n=70 for the high volume dose because 7 subjects titrated up from the 40 IU/kg arm and will be displayed in both arms.
Arm/Group | CSL830 (40) | CSL830 (60)
Number analyzed (Participants) | 63 | 70
events/year
  AEs Leading to Premature Study Discontinuation | 0.01 | 0.03
  Thromboembolic Events | 0.00 | 0.01
  Anaphylaxis | 0.00 | 0.00
  HAE Attacks Resulting in In-Patient Hospitalizatio | 0.00 | 0.00
  Solicited AEs Graded as Severe | 0.00 | 0.00
  Related SAEs Other Than Specified Above | 0.00 | 0.00
  Antibodies to C1-INH (Inhibitory + Non-inhibitory) | 0.06 | 0.09

3. Secondary Outcome: Percentage of Subjects Who Have Solicited Adverse Events (AEs)
Description: The number of subjects having at least 1 solicited local AE during a treatment were divided by the number of subjects in the corresponding treatment. The analysis population for this endpoint was the Safety Population: The Safety Population comprised all subjects who provided informed consent / assent, who were randomized, and who received at least 1 dose or a partial dose of CSL830.
Time Frame: Up to 146 weeks
Population: as for outcome 1
Measure: Number; unit: Percent of subjects
Groups:
- CSL830 (60): A high-volume dose of C1-INH (60 IU/kg) administered subcutaneously twice a week. Note: Actual n=70 for the high volume dose because 7 subjects titrated up from the 40 IU/kg arm and will be displayed in both arms.
Arm/Group | CSL830 (40) | CSL830 (60)
Number analyzed (Participants) | 63 | 70
Percent of subjects | 55.6 | 45.7

4. Secondary Outcome: Percentage of Injections Followed by At Least One Solicited Adverse Event
Description: The percent of injections followed by at least one solicited adverse event. The analysis population for this endpoint was the Safety Population: The Safety Population comprised all subjects who provided informed consent / assent, who were randomized, and who received at least 1 dose or a partial dose of CSL830. This was assessed across all participants, calculated as total number of events following injections / total number of injections across all participants, in each Arm.
Time Frame: Up to 146 weeks
Population: as for outcome 1
Measure: Number; unit: Percent of injections
Groups:
- CSL830 (60): A high-volume dose of C1-INH (60 IU/kg) administered subcutaneously twice a week. Actual n= 70 because 7 subjects titrated up from the 40IU/kg arm and will be displayed in both arms.
Arm/Group | CSL830 (40) | CSL830 (60)
Number analyzed (Participants) | 63 | 70
Percent of injections | 6.3 | 5.1

5. Secondary Outcome: Percentage of Subjects Who Become Seropositive for Human Immunodeficiency Virus (HIV-1/-2), Hepatitis B Virus, or Hepatitis C Virus.
Description: Blood samples to be tested for HIV-1/-2, HBV, and HCV. The analysis population for this endpoint was the Safety Population: The Safety Population comprised all subjects who provided informed consent / assent, who were randomized, and who received at least 1 dose or a partial dose of CSL830.
Time Frame: Up to 146 weeks
Population: as for outcome 1
Measure: Number; unit: Percent of Subjects
Arm/Group | CSL830 (40) | CSL830 (60)
Number analyzed (Participants) | 63 | 70
Percent of Subjects | 0 | 0

6. Secondary Outcome: Percentage of Subjects Who Experience a Time-normalized HAE Attack Frequency of <1 HAE Attack Per 4-Week Period
Description: The percentage of subjects with a time-normalized merged HAE attack frequency of <1 HAE attack per 4-week period. The analysis population for this endpoint was the Intent-to-Treat (ITT) Population: The ITT Population comprised all subjects who provided informed consent / assent and were randomized, regardless of whether or not they received CSL 830.
Time Frame: Up to 146 weeks
Population: Intent-to-Treat (ITT) Population: The ITT Population comprised all subjects who provided informed consent / assent and were randomized, regardless of whether or not they received CSL 830.
Measure: Number; unit: Percent of Subjects
Arm/Group | CSL830 (40) | CSL830 (60)
Number analyzed (Participants) | 63 | 63
Percent of Subjects | 79.4 | 85.7

7. Secondary Outcome: Percentage of Subjects Who Are Responders
Description: A responder was defined as a subject with a ≥ 50% reduction in the time-normalized number of HAE attacks on CSL830 relative to the time-normalized number of HAE attacks used to qualify for participation in the current study. The analysis population for this endpoint was the Intent-to-Treat (ITT) Population: The ITT Population comprised all subjects who provided informed consent / assent and were randomized, regardless of whether or not they received CSL830. Not all subjects in the ITT were available for this outcome measure.
Time Frame: Up to 146 weeks
Population: Intent-to-Treat (ITT) Population: The ITT Population comprised all subjects who provided informed consent / assent and were randomized, regardless of whether or not they received CSL830.
Measure: Number (95% Confidence Interval); unit: Percent of Subjects
Arm/Group | CSL830 (40) | CSL830 (60)
Number analyzed (Participants) | 62 | 60
Percent of Subjects | 93.5 [84.6 to 97.5] | 91.7 [81.9 to 96.4]

ADVERSE EVENTS:
Time Frame: 146 weeks per subject
Description: n=70 because 7 subjects titrated up from the 40 IU/kg arm and will be displayed in both arms.
Arm/Group | CSL830 (40) | CSL830 (60)
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/70
Serious Adverse Events (participants affected / at risk) | 4/63 | 5/70
Other Adverse Events (participants affected / at risk) | 33/63 | 28/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSL830 (40) (N=63) | CSL830 (60) (N=70)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSL830 (40) (N=63) | CSL830 (60) (N=70)
Contusion (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Headache (Nervous system disorders) | 10 (22) | 10 (19)
Migraine (Nervous system disorders) | 4 (8) | 0 (0)
Injection site pain (General disorders) | 17 (211) | 10 (51)
Injection site erythema (General disorders) | 10 (45) | 12 (331)
Injection site bruising (General disorders) | 9 (56) | 7 (22)
Injection site reaction (General disorders) | 5 (75) | 8 (72)
Injection site haematoma (General disorders) | 6 (11) | 4 (12)
Injection site induration (General disorders) | 4 (19) | 3 (4)
Injection site swelling (General disorders) | 4 (19) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (10) | 4 (14)
Diarrhoea (Gastrointestinal disorders) | 4 (12) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 1 (6)
Nasopharyngitis (Infections and infestations) | 12 (23) | 21 (36)
Upper respiratory tract infection (Infections and infestations) | 8 (10) | 8 (10)
Urinary tract infection (Infections and infestations) | 3 (4) | 6 (6)
Bronchitis (Infections and infestations) | 7 (7) | 2 (2)
Sinusitis (Infections and infestations) | 4 (4) | 4 (7)

LIMITATIONS AND CAVEATS:
None reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-07-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT02316353/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT02316353/SAP_001.pdf